CLINICAL TRIAL: NCT00961298
Title: An Open Label Trial of Duloxetine in the Treatment of Irritable Bowel Syndrome and Comorbid Generalized Anxiety Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: West Penn Allegheny Health System (Other)
Responsible Party: Principal Investigator, Alicia Kaplan, MD, West Penn Allegheny Health System
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: RC-4656
Record Dates: First submitted 2009-08-17; First posted 2009-08-18 (Estimated); Results first posted 2014-07-09 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-06

CONDITIONS: Irritable Bowel Syndrome; Generalized Anxiety Disorder
Keywords: IBS; Irritable Bowel Syndrome; GAD; Generalized Anxiety Disorder
MeSH Terms: conditions — Irritable Bowel Syndrome; Generalized Anxiety Disorder | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Duloxetine (Experimental): Two weeks of placebo run in followed by 12 weeks of Duloxetine.
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: Duloxetine — All subjects will receive single-blind placebo for the first two weeks, and then duloxetine for the next 12 weeks, followed by an up to 2 week taper off of the duloxetine. After 2 weeks of placebo daily, subjects will receive 30 mg per day of duloxetine for two weeks, then titrated up to 60 mg per day of duloxetine at week 2. A dosage decrease to 30 mg daily is permittable after week 2. This will be a flexible dose study with doses of duloxetine progressively increasing at weeks 4 (90 mg daily) and 6 (120 mg daily) in conjunction with CGI-I scores, to reach 120 mg daily or the maximum tolerated dose, if less than 120 mg daily at Week 12. There will be a post-taper follow up appointment at Week 14. Of Note: Amendment IRB Approved 6/14/11 Study Ending at Week 12 with removal of Week 14 visit as part of study.
  Other Names: Cymbalta

SUMMARY:
The investigators propose to evaluate the effectiveness of duloxetine in treating subjects with both Irritable Bowel Syndrome (IBS) and Generalized Anxiety Disorder (GAD). The investigators hypothesize that duloxetine as a single therapeutic agent will effectively target pain and other core symptoms of IBS as well as GAD in this patient population with both conditions.

DETAILED DESCRIPTION:
Generalized Anxiety Disorder (GAD) is commonly associated with Irritable Bowel Syndrome(IBS). The etiology of IBS remains unknown and it is often refractory to treatment. Duloxetine has demonstrated efficacy in the treatment of GAD as well as other pain disorders including fibromyalgia and diabetic neuropathy.

We plan to study 30 subjects with diagnoses of IBS and GAD between the ages of 18 and 65 years. There will be a single-blind placebo-run-in for the first 2 weeks, followed by open-label duloxetine for 12 weeks flexibly titrated to 120 mg/day. Subjects will be informed that they will receive placebo for 2 weeks during the trial. All study visits will be at Allegheny General Hospital Department of Psychiatry. The study consists of a total of nine office visits.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* Active IBS diagnosis by a gastroenterologist
* Generalized Anxiety Disorder diagnosed by DSM-IV TR criteria and the Mini International Neuropsychiatric Interview for the DSM-IV (Mini)
* No changes in any non study medication once starting the study

Exclusion Criteria:

* Current diagnoses of Major Depressive Disorder, Panic Disorder, Social Phobia, Post Traumatic Stress Disorder, Obsessive Compulsive Disorders, Eating Disorders, Somatoform Disorders, Drug or alcohol abuse or dependence, or severe personality disorder
* Lifetime history of any Bipolar Disorder or Psychotic Disorder
* Concurrent GI disorders falling outside of Rome III Functional GI disorders
* Pregnant women or sexually active female subjects not using medically acceptable method of contraception
* Current suicidal ideation
* Unstable medical condition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alicia J Kaplan, MD, Principal Investigator — West Penn Allegheny Health System

REFERENCES:
- [Derived] Kaplan A, Franzen MD, Nickell PV, Ransom D, Lebovitz PJ. An open-label trial of duloxetine in patients with irritable bowel syndrome and comorbid generalized anxiety disorder. Int J Psychiatry Clin Pract. 2014 Jan;18(1):11-5. doi: 10.3109/13651501.2013.838632. Epub 2013 Sep 20. PMID 23980534

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were referred by a gastroenterologist who had Irritable Bowel Syndrome and anxiety.
Pre-assignment Details: Two participants were considered screen failures and were not entered into the placebo run in phase.
Groups:
- Treatment Arm: Every study eligible subject entered a two week placebo run in followed by 12 weeks treatment intervention with Duloxetine.
Period: Two Week Placebo Run in
Arm/Group | Treatment Arm
Started | 15
Completed | 14
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: 12 Weeks Duloxetine Treatment Phase
Arm/Group | Treatment Arm
Started | 14
Completed | 11
Not Completed | 3
Not completed — Withdrawal by Subject | 2
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Groups:
- Treatment Arm: every subject had a two week placebo run in followed by 12 weeks treatment intervention with Duloxetine.
Arm/Group | Treatment Arm
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.54 (12.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Clinical Global Impression Scale
Description: The scale consists of two parts the first part being Severity of Illness and the second part is Global Improvement. We report the Global improvement scale.
  The Global Improvement is a 1-7 change scale of global improvement since inclusion in the project ranging with 1 "very much improved", 4 "no change", and 7 "very much worse."
Time Frame: endpoint [12 weeks]
Population: per protocol
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- Treatment Arm: every study eligible subject had a two week placebo run in followed by 12 weeks treatment intervention with Duloxetine.
Arm/Group | Treatment Arm
Number analyzed (Participants) | 11
scores on a scale | 2.64 (0.5)

2. Secondary Outcome: Hamilton Anxiety Rating Scale
Description: The HAM-A is a 14 question scale with five responses. Responses range from 0 "not present" to 4 "very severe." The total score ranges from 0 to 56. Higher values represent a worse outcome.
Time Frame: endpoint [12 weeks]
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Treatment Arm
Number analyzed (Participants) | 11
scores on a scale | 9.75 (4.5)

3. Secondary Outcome: Irritable Bowel Syndrome-Quality of Life Scale
Description: The IBS-QOL consists of 34 items, each with a five-point response scale. Ratings range from 1 "not at all" to 5 "extremely" or "a great deal" Higher responses on the scale indicate worse outcome. A minimal total score would be 34, maximum 170.
Time Frame: endpoint [12 weeks]
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Treatment Arm
Number analyzed (Participants) | 11
scores on a scale | 81.73 (19.25)

4. Secondary Outcome: Irritable Bowel Syndrome Severity Scoring System
Description: This is a 4 item Likert scale with each assessment being 100 mm scored from measuring from 0 to 400. Higher numbers indicate worse outcome.
Time Frame: endpoint [12 weeks]
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Treatment Arm
Number analyzed (Participants) | 11
scores on a scale | 187.09 (54.05)

ADVERSE EVENTS:
Time Frame: within 14 weeks.
Description: patient interview at study visit.
Arm/Group | Treatment Arm
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 9/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=15)
constipation (Gastrointestinal disorders) | 3 (3)
nausea (Gastrointestinal disorders) | 5 (5)
fatigue (General disorders) | 5 (5)
dry mouth (Gastrointestinal disorders) | 1 (1)
anxiety (Psychiatric disorders) | 1 (1)
dizziness (Nervous system disorders) | 3 (3)
weight gain (Endocrine disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
A limitation of this pilot study was its small sample size and open label design. Another limitation may be that the patient sample is not representative of a true cross section of the GAD population as a whole.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No